CLINICAL TRIAL: NCT00334035
Title: Duration of Maintenance Anti-psychotic Therapy After First -Episode Schizophrenia: a Double-blind Randomized Placebo-control Relapse Prevention Study
Brief Title: Antipsychotic Therapy and First Episode
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: D1441C09906
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2008-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
For schizophrenic patients who remained in remission while on maintenance medication, there may come a point in time when the relative risk for relapse become so low that discontinuation of therapy can be considered. This study is to investigate whether that point in time is reached in 12 months following the first episode illness. Moreover, it also aims to identify other predictors of relapse as well as to evaluate the costs and benefits of maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, from 18 to 65 years of age at Visit 1
* Patients must achieve a level of understanding and expressive capacity sufficient to communicate adequately with the study coordinator and to participate in cognitive testing.
* Patients must agree to cooperate with all tests and examinations required by the protocol. They must be willing to comply fully with treatment
* Patient must understand the nature of the study and must sign an informed consent document.
* Patients must be Cantonese speaking Han Chinese
* Patients must be diagnosed, according to the SCID for DSM-IV, with schizophrenia, schizoaffective disorder or schizophreniform psychosis.
* Patients must have good response to anti-psychotic treatment by achieving a rating of 2 or below in Clinical Global Impression Scale (CGI) Severity of illness; a rating of 4 or below in Improvement scale, and a rating of 3 or below in (conceptual disorganization, unusual thought content), a rating of 2 or below in (delusion, hallucinatory behavior) and a rating of 4 or below in (Suspiciousness) of Positive and Negative Syndrome Scale (PANSS) for at least 8 weeks

Exclusion Criteria:

* Female patients who are either pregnant or lactating.
* Patients previously on clozapine should be excluded from the study
* Significant medical illnesses including seizures.
* DSM-IV substance (alcohol or other drugs) abuse or dependence within the past 3 months.
* Judged clinically to be at serious suicidal risk.
* Treatment with an injectable depot neuroleptic within less than one of the patient's dosing intervals between depot neuroleptic injections prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2003-08; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
For patients in remission while on maintenance medication, the study investigates whether medication discontinuation can be reached in 12 months following a first episode illness.

SECONDARY OUTCOMES:
Predictors of relapse, and costs and benefits of maintenance therapy in terms of functioning, quality of life, side effects, carer's burden, negative symptoms and cognitive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eric YH Chen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Research Site, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Hui CLM, Honer WG, Lee EHM, Chang WC, Chan SKW, Chen ESM, Pang EPF, Lui SSY, Chung DWS, Yeung WS, Ng RMK, Lo WTL, Jones PB, Sham P, Chen EYH. Long-term effects of discontinuation from antipsychotic maintenance following first-episode schizophrenia and related disorders: a 10 year follow-up of a randomised, double-blind trial. Lancet Psychiatry. 2018 May;5(5):432-442. doi: 10.1016/S2215-0366(18)30090-7. Epub 2018 Mar 15. PMID 29551618
- [Derived] Chen EY, Hui CL, Lam MM, Chiu CP, Law CW, Chung DW, Tso S, Pang EP, Chan KT, Wong YC, Mo FY, Chan KP, Yao TJ, Hung SF, Honer WG. Maintenance treatment with quetiapine versus discontinuation after one year of treatment in patients with remitted first episode psychosis: randomised controlled trial. BMJ. 2010 Aug 19;341:c4024. doi: 10.1136/bmj.c4024. PMID 20724402